CLINICAL TRIAL: NCT01352715
Title: Multicenter Study of Options for Second-Line Effective Combination Therapy (SELECT)
Brief Title: Study of Options for Second-Line Effective Combination Therapy (SELECT)
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5273; 1U01AI068636 (NIH); 5UM1AI068634 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-05-12 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Lopinavir; lopinavir-ritonavir drug combination; Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine, and zidovudine drug combination; abacavir, lamivudine drug combination; lamivudine, zidovudine drug combination; abacavir; Zidovudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: LPV/r plus RAL (Experimental): Participants were administered LPV/r plus RAL orally twice daily throughout follow-up.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Raltegravir
- Arm B: LPV/r plus best available NRTIs (Experimental): Participants were administered LPV/r orally twice daily, plus NRTI options provided by the study, to include the best available NRTIs (listed below) throughout follow-up-
  * FTC/TDF orally twice daily
  * ABC/3TC/ZDV orally twice daily
  * ABC/3TC orally once daily
  * 3TC/ZDV orally twice daily
  * ABC 300mg orally twice daily or 600 mg once daily
  * 3TC orally twice daily
  * ZDV orally twice daily
  Interventions: Drug: Lopinavir/ritonavir; Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Abacavir/lamivudine/zidovudine; Drug: Abacavir/lamivudine; Drug: Lamivudine/zidovudine; Drug: Abacavir; Drug: Zidovudine; Drug: Lamivudine

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Lopinavir 400mg/ritonavir 100mg (given as two LPV 200mg/RTV 50mg fixed-dose combination tablets) orally twice daily, with or without food, throughout follow-up.
  Other Names: Aluvia; LPV/r; Kaletra
Drug: Lopinavir/ritonavir — Lopinavir 400mg/ritonavir 100mg (given as three LPV 133.3 mg/RTV 33.3 mg fixed-dose combination soft gelatin capsules) orally twice daily, with food, throughout follow-up.
  Other Names: Kaletra; LPV/r
Drug: Raltegravir — Raltegravir 400 mg tablet orally twice daily, with or without food, throughout follow-up.
  Other Names: Isentress; RAL
  Arms: Arm A: LPV/r plus RAL
Drug: Emtricitabine/tenofovir disoproxil fumarate — Emtricitabine 200 mg/tenofovir disoproxil fumarate 300mg fixed-dose combination tablet orally once daily, with or without food, throughout follow-up.
  Other Names: Truvada; FTC/TDF
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Abacavir/lamivudine/zidovudine — Abacavir 300 mg/lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily, with or without food, throughout follow-up.
  Other Names: Trizivir; ABC/3TC/ZDV
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Abacavir/lamivudine — Abacavir 600 mg/lamivudine 300 mg fixed-dose combination tablet orally once daily, with or without food, throughout follow-up.
  Other Names: Epzicom; ABC/3TC
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Lamivudine/zidovudine — Lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily, with or without food, throughout follow-up.
  Other Names: Combivir; CBV; 3TC/ZDV
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Abacavir — Abacavir 300 mg tablet orally twice daily or 600 mg (given as two 300 mg tablets) once daily, with or without food, throughout follow-up.
  Other Names: Ziagen; ABC
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Zidovudine — Zidovudine 300 mg tablet orally twice daily, with or without food, throughout follow-up.
  Other Names: Retrovir; ZDV
  Arms: Arm B: LPV/r plus best available NRTIs
Drug: Lamivudine — Lamivudine 150 mg tablet orally twice daily, with or without food, throughout follow-up.
  Other Names: Epivir; 3TC
  Arms: Arm B: LPV/r plus best available NRTIs

SUMMARY:
The study was conducted on people who were taking their first anti-HIV drug regimen (including an Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI), a type of anti-HIV drug) but the drugs in this regimen were not doing a good job of fighting their HIV infection.

The main purpose of this study was to compare two other anti-HIV drug regimens to see how well they fight HIV. The study also looked at how well participants tolerate the drug regimens and how safe they are.

The study was designed to determine whether taking the combination of lopinavir/ritonavir (LPV/r) plus raltegravir (RAL) works as well as what is usually used for second-line therapy: LPV/r plus the best-available nucleoside (nucleotide) reverse transcriptase inhibitor (NRTI) combination. Testing a regimen that does not include any NRTIs was important because NRTIs may no longer work for patients who received them as part of their first treatment regimen.

DETAILED DESCRIPTION:
As more HIV-infected persons start antiretroviral therapy (ART) worldwide, the number needing second-line therapy is increasing. In many settings, an NNRTI-based regimen is the preferred first-line ART, whereas a protease inhibitor (PI)-based regimen is often reserved for second-line ART. Both of these types of regimens usually include two NRTIs.

As with initial ART, second-line regimens ideally should be composed of three fully active drugs that have potent anti-HIV activity to maximize the chances of durable viral suppression. However, such a goal may not be achieved with second-line PI-based regimens containing NRTIs because of resistance mutations from first-line therapy that reduce the activity of the NRTI class. The most significant of these mutations include M184V, thymidine analogue mutations (TAMs), Q151M complex, and K65R. The presence of K65R would result in resistance to most NRTIs (leaving only zidovudine (ZDV) and possibly abacavir (ABC) as active second-line options); the presence of multiple TAMs and/or Q151M alone or in complex with other mutations would also result in resistance to most NRTIs.

Recent data suggest that patients with isolated M184V-related NRTI resistance who subsequently switch to a boosted PI plus lamivudine (3TC)- or emtricitabine (FTC)-based regimen may achieve HIV-1 RNA suppression without the need to switch to more complex regimens [1]. Detection of an isolated M184V NRTI mutation is possible when resources allow for early diagnosis of virologic failure. However, in many resource-limited settings (RLS) early diagnosis of virologic failure is difficult because of infrequent monitoring of viral load or unavailability of viral load testing. This study intended to provide information applicable to the vast majority of RLS where resistance testing is not used routinely for selection of second-line regimens and PIs not needing refrigeration are preferred.

This was a phase III, dual-arm, open-label, randomized, non-inferiority study for participants who were on a failing NNRTI-containing first-line regimen. The study evaluated the difference in virologic failure rate between two treatment arms:

Arm A: LPV/r plus RAL Arm B: LPV/r plus best available NRTIs

Best available NRTI combinations were selected by the site investigator prior to randomization from a list of combinations approved by the study or in consultation with the A5273 Clinical Management Committee (CMC). The NRTIs provided by the study were FTC/TDF, ABC/3TC/ZDV, ABC/3TC, 3TC/ZDV, ABC, 3TC, and ZDV.

Participants took their assigned study therapy until 96 weeks of follow-up or 52 weeks after the last participant was enrolled (protocol amendment), whichever was earlier. This study originally planned to enroll 600 participants (300 per study arm), but the sample size was re-evaluated to 480 participants (240 per study arm), due to emergent data from other studies. Participants were assigned with equal probability to one of the two treatment regimens using permuted blocks. Randomization was stratified by three factors: screening HIV-1 RNA (≥100,000 versus <100,000 copies/mL); screening CD4+ cell count (≥100 versus <100 cells/mm3), and selection of ZDV in the NRTI regimen (yes/no). Furthermore, randomization was balanced by site.

During the study, participants were asked to return to the clinic at Weeks 4, 12, 24, and then every 12 weeks. Visits lasted about 30 minutes. At most visits, participants had a physical exam, had their arm, waist and hip circumference measured, and answered questions about their medical condition and any medications they were taking. At some visits, participants completed questionnaires to see how they were feeling, if they had been hospitalized recently, and how well they were taking their anti-HIV drugs, had their blood drawn and were asked to give urine samples. If the participant was female and able to become pregnant, a pregnancy test was taken at any visit that pregnancy was suspected.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Confirmation of first-line virologic failure
* Certain laboratory values obtained within 45 days prior to study entry. More information on this criterion can be found in the study protocol.
* Negative pregnancy test within 48 hours prior to study entry.
* Must refrain from participating in a conception process, and, if participating in sexual activity that could lead to pregnancy, must use at least one acceptable type of contraceptive. More information on this criterion can be found in the study protocol.
* Karnofsky performance score >= 70 within 45 days prior to study entry.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* No intention to relocate away from current geographical area of residence for the duration of study participation.

Exclusion Criteria:

* Use of any immunomodulator, HIV vaccine, or other investigational therapy within 45 days prior to study entry, with the exception of a tapering course of corticosteroids as acute therapy for pneumocystis jiroveci pneumonia (PCP) or acute asthma/chronic obstructive pulmonary disease flare and/or prednisone at a daily dose of <10 mg (physiologic replacement dose).
* If the potential participant has had resistance testing, evidence of broad NRTI cross-resistance that, in the opinion of the investigator, would not allow selection of an effective NRTI combination if the participant were randomized to the LPV/r + best available NRTIs arm.
* Prior exposure to a Protease Inhibitor.
* Known history of congenital long QT syndrome, hypokalemia, or planned use of other drugs that prolong the QT interval.
* Pregnancy or breast-feeding.
* Known history of chronic hepatitis B virus (HBV) infection or current HBV infection defined by the presence of hepatitis B surface antigen in serum or plasma.
* Active tuberculosis (TB) requiring treatment with rifampicin.
* Previously diagnosed malignancies other than basal cell carcinoma and cutaneous Kaposi sarcoma.
* Requirement for taking any medications that are prohibited with the study drugs. More information on this criterion can be found in the study protocol, section 5.4.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Active drug or alcohol use or dependence or other condition that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2014-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M La Rosa, MD, Study Chair — Asociacion Civil Impacta Salud y Educacion - Miraflores, CRS; Ann C Collier, MD, Study Chair — Univ. of Washington Clinical HIV Research Program (CHIRP)
Locations (16):
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- India (3):
  - BJ Medical College CRS (31441), Pune, Maharashtra
  - NARI Pune CRS, Pune, Maharashtra
  - Y.R.G Ctr, for AIDS Research and Education (11701), Chennai
- AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS (12601), Eldoret, Kenya
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe CRS (12001), Lilongwe
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Barranco CRS (11301), Lima
- South Africa (4):
  - Wits HIV CRS (11101), Johannesburg, Gauteng
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
  - Univ. of Witwatersrand CRS (11101), Johannesburg
- Kilimanjaro Christian Medical CRS, Kilimanjaro Region, Moshi, Tanzania
- Chiang Mai University ACTG CRS (11501), Chiang Mai, Thailand
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Background] [1] Hull M, Moore D, Harris M, et al. A lamivudine (3TC)-based backbone in conjunction with a boosted protease inhibitor (PI) is sufficient to achieve virologic suppression in the presence of M184V mutations. Program and abstracts of the 49th Interscience Conference on Antimicrobial Agents and Chemotherapy; September 12-15, 2009; San Francisco, California. Abstract H-916.
- [Derived] Torres TS, Harrison LJ, La Rosa AM, Zheng L, Cardoso SW, Ulaya G, Akoojee N, Kadam D, Collier AC, Hughes MD; for AIDS Clinical Trials Group (ACTG) A5273 Study Group. Poor quality of life and incomplete self-reported adherence predict second-line ART virological failure in resource-limited settings. AIDS Care. 2021 Oct;33(10):1340-1349. doi: 10.1080/09540121.2021.1874275. Epub 2021 Jan 23. PMID 33487029
- [Derived] La Rosa AM, Harrison LJ, Taiwo B, Wallis CL, Zheng L, Kim P, Kumarasamy N, Hosseinipour MC, Jarocki B, Mellors JW, Collier AC; ACTG A5273 Study Group. Raltegravir in second-line antiretroviral therapy in resource-limited settings (SELECT): a randomised, phase 3, non-inferiority study. Lancet HIV. 2016 Jun;3(6):e247-58. doi: 10.1016/S2352-3018(16)30011-X. Epub 2016 Apr 18. PMID 27240787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at international AIDS Clinical Trials Group Units. Recruitment occurred between March 13, 2012 (date first participant was randomized) and October 2, 2013 (date last participant was randomized).
Pre-assignment Details: 515 were randomized 1:1 to treatment arms A and B.
Groups:
- Arm A: LPV/r Plus RAL: Participants were administered LPV/r plus RAL orally twice daily.
  Lopinavir/ritonavir: Lopinavir 400mg/ritonavir 100mg orally twice daily.
  Raltegravir: Raltegravir 400 mg tablet orally twice daily.
- Arm B: LPV/r Plus Best Available NRTIs: Participants were administered LPV/r orally twice daily, plus NRTI options provided by the study, to include the best available NRTIs.
  Lopinavir/ritonavir: Lopinavir 400mg/ritonavir 100mg orally twice daily.
  Emtricitabine/tenofovir disoproxil fumarate: Emtricitabine 200 mg/tenofovir disoproxil fumarate 300mg fixed-dose combination tablet orally once daily.
  Abacavir/lamivudine/zidovudine: Abacavir 300 mg/lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily.
  Abacavir/lamivudine: Abacavir 600 mg/lamivudine 300 mg fixed-dose combination tablet orally once daily.
  Lamivudine/zidovudine: Lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily.
  Abacavir: Abacavir 300 mg tablet orally twice daily or 600 mg (given as two 300 mg tablets) once daily.
  Zidovudine: Zidovudine 300 mg tablet orally twice daily.
  Lamivudine: Lamivudine 150 mg tablet orally twice daily.
Period: Overall Study
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Started | 260 | 255
Completed | 215 | 209
Not Completed | 45 | 46
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 4 | 8
Not completed — site closure | 16 | 15
Not completed — no final visit in closeout period | 15 | 12
Not completed — major ineligibility | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat: All 512 participants without a major eligibility violation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs | Total
Number analyzed (Participants) | 258 | 254 | 512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 258 | 254 | 512
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (8) | 38 (8) | 39 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 126 | 260
  Male | 124 | 128 | 252
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 0 | 1 | 1
  Black Non-Hispanic | 164 | 162 | 326
  Hispanic (Regardless of Race) | 11 | 9 | 20
  Asian, Pacific Islander | 83 | 82 | 165
Region of Enrollment [Number; unit: participants]
  Malawi | 56 | 55 | 111
  South Africa | 52 | 51 | 103
  India | 80 | 78 | 158
  Zimbabwe | 24 | 23 | 47
  Kenya | 24 | 24 | 48
  Peru | 5 | 4 | 9
  Brazil | 6 | 6 | 12
  Tanzania | 8 | 9 | 17
  Thailand | 3 | 4 | 7
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.6 (0.8) | 4.5 (0.9) | 4.5 (0.8)
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/mm^3] | 178 (170) | 182 (160) | 180 (165)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Virologic Failure by Week 48
Description: The primary endpoint was time to virologic failure. Virologic failure was defined as confirmed viral load >400 copies/mL at or after week 24. The Kaplan-Meier estimate of the cumulative probability of virologic failure by week 48 was used.
Time Frame: From study entry to week 48
Population: Intention to treat: All 512 participants without a major eligibility violation were included in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 254
cumulative probability per 100 persons | 10.3 [6.5 to 14.0] | 12.4 [8.3 to 16.5]
Statistical Analysis 1: Comparison: Arm A: LPV/r Plus RAL vs Arm B: LPV/r Plus Best Available NRTIs; Treatment comparison was made using the difference (arm A - arm B) in the stratified Kaplan-Meier estimate for the week 48 cumulative probability of virologic failure with 95% confidence interval; Test type: Non-Inferiority or Equivalence — Confidence interval estimation was stratified by randomization stratification factors using Greenwood's variance with the inverse of this variance used for the stratum weights. The pre-specified upper confidence bound for non-inferiority was 10 percentage points; Cumulative probability difference = -3.4, 95% CI 2-sided [-8.4 to 1.5]

2. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 48
Description: Change in CD4+ cell count was calculated as CD4+ cell count at week 48 minus CD4+ cell count at study entry.
Time Frame: Study entry and week 48
Population: Intention to treat: All 488 participants without a major eligibility violation, and with baseline and week 48 data available were used in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 246 | 242
cells/mm^3 | 199 [181 to 218] | 190 [171 to 209]

3. Secondary Outcome: Number of Participants With HIV-1 Drug Resistance Mutations in Protease, Reverse Transcriptase, and Integrase in Participants With Virologic Failure at Baseline and at Time of Virologic Failure
Description: Mutations were defined as major IAS mutations in the IAS-USA July 2014 list. New mutations were those detected at virologic failure but not at baseline.
Time Frame: From study entry through to week 96
Population: Participants with virologic failure, and with a pair of baseline and virologic failure sequences available, were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 39 | 45
participants
  No new IAS mutations | 29 | 32
  1-2 new IAS mutations | 9 | 13
  3 new IAS mutations | 1 | 0

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Event (AE) at Least One Grade Higher Than Baseline
Description: The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs.
Time Frame: From start of randomized treatment to off randomized treatment (up to 96 weeks)
Population: As treated: Participants on randomized treatment are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 253
participants | 62 | 81

5. Secondary Outcome: Number of Participants Discontinuing Randomized Treatment for Toxicity
Description: Discontinuation of randomized treatment for toxicity included participant decision to discontinue for low grade toxicity. Within class NRTI changes were not considered discontinuations.
Time Frame: From Start of Randomized Treatment to Off Randomized Treatment (up to 96 weeks)
Population: Competing risk approach: Time was measured from start of randomized treatment until the date of randomized treatment discontinuation for toxicity. Randomized treatment discontinuation for other reasons was considered as an independent competing risk, and participants discontinuing the study were censored on the date of last participant contact.
Measure: Number; unit: participants
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 253
participants | 3 | 3

6. Secondary Outcome: Number of Participants With a New AIDS-defining Events or Death
Description: AIDS-defining events were those recognized by the Centers for Disease Control (CDC) and World Health Organization (WHO)
Time Frame: From study entry throughout follow-up (up to 96 weeks)
Population: Intention to treat: All 512 participants without major eligibility violations were in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Number; unit: participants
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 254
participants | 15 | 17

7. Secondary Outcome: Number of Participants With a Targeted Serious Non-AIDS-defining Event or Death
Description: Serious non-AIDS diagnoses were based on ACTG Appendix 60 Diagnosis Codes
Time Frame: From study entry throughout follow-up (up to 96 weeks)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 254
participants | 7 | 7

8. Secondary Outcome: Percentage of Time Spent in Hospital
Description: The percentage of total study time that participants were in hospital.
Time Frame: From study entry throughout follow-up (up to 96 weeks)
Population: Intention to treat: All 512 participants without a major eligibility violation were in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Number; unit: percentage of time spent in hospital
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 254
percentage of time spent in hospital | 0.08 | 0.12

9. Secondary Outcome: Changes in Fasting Total Cholesterol, High-density Lipoprotein (HDL) Cholesterol, Low-density Lipoprotein (LDL) Cholesterol, Triglycerides, and Glucose From Baseline
Description: Fasting was for 8 hours and the metabolic panel was drawn locally.
Time Frame: Study entry and week 48
Population: Intention to treat: All 512 participants without a major eligibility violation with data available at entry and week 48 were included in their assigned randomized treatment arm. total cholesterol (Arm A N=216 B N=220) HDL (Arm A N=219 B N=223) LDL (Arm A N=202 B N=205) triglycerides (Arm A N=219 B N=222), glucose (Arm A N=213 B N=223)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: LPV/r Plus RAL | Arm B: LPV/r Plus Best Available NRTIs
Number analyzed (Participants) | 258 | 254
mg/dL
  total cholesterol change | 31 [24 to 38] | 15 [9 to 20]
  high-density lipoprotein (HDL) cholesterol change | 4 [2 to 6] | 2 [0 to 4]
  low-density lipoprotein (LDL) cholesterol change | 17 [12 to 21] | 10 [6 to 15]
  triglycerides change | 80 [51 to 109] | 31 [13 to 49]
  glucose change | 2 [0 to 5] | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: From study entry throughout follow-up (up to 96 weeks)
Description: The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs. Expedited adverse event reporting followed "Manual for Expedited Reporting of Adverse Events to DAIDS" (DAIDS EAE Manual), version 2.0 January, 2010.
Groups:
- LPV/r + RAL: Participants were administered LPV/r plus RAL orally twice daily. Lopinavir/ritonavir: Lopinavir 400mg/ritonavir 100mg orally twice daily. Raltegravir: Raltegravir 400 mg tablet orally twice daily.
- LPV/r + NRTIs: Participants were administered LPV/r orally twice daily, plus NRTI options provided by the study, to include the best available NRTIs.
  Lopinavir/ritonavir: Lopinavir 400mg/ritonavir 100mg orally twice daily. Emtricitabine/tenofovir disoproxil fumarate: Emtricitabine 200 mg/tenofovir disoproxil fumarate 300mg fixed-dose combination tablet orally once daily.
  Abacavir/lamivudine/zidovudine: Abacavir 300 mg/lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily.
  Abacavir/lamivudine: Abacavir 600 mg/lamivudine 300 mg fixed-dose combination tablet orally once daily.
  Lamivudine/zidovudine: Lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet orally twice daily.
  Abacavir: Abacavir 300 mg tablet orally twice daily or 600 mg (given as two 300 mg tablets) once daily.
  Zidovudine: Zidovudine 300 mg tablet orally twice daily. Lamivudine: Lamivudine 150 mg tablet orally twice daily.
Arm/Group | LPV/r + RAL | LPV/r + NRTIs
Serious Adverse Events (participants affected / at risk) | 19/258 | 30/254
Other Adverse Events (participants affected / at risk) | 252/258 | 250/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r + RAL (N=258) | LPV/r + NRTIs (N=254)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Toxic optic neuropathy (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
AIDS dementia complex (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Leptospirosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r + RAL (N=258) | LPV/r + NRTIs (N=254)
Diarrhoea (Gastrointestinal disorders) | 16 | 25
Vomiting (Gastrointestinal disorders) | 7 | 13
Pyrexia (General disorders) | 22 | 23
Oral candidiasis (Infections and infestations) | 15 | 12
Upper respiratory tract infection (Infections and infestations) | 19 | 16
Urinary tract infection (Infections and infestations) | 13 | 13
Alanine aminotransferase increased (Investigations) | 55 | 40
Aspartate aminotransferase increased (Investigations) | 70 | 61
Blood alkaline phosphatase increased (Investigations) | 67 | 73
Blood bicarbonate decreased (Investigations) | 79 | 85
Blood bilirubin increased (Investigations) | 27 | 16
Blood calcium decreased (Investigations) | 38 | 40
Blood cholesterol increased (Investigations) | 150 | 121
Blood creatinine increased (Investigations) | 9 | 17
Blood glucose decreased (Investigations) | 15 | 13
Blood glucose increased (Investigations) | 40 | 36
Blood phosphorus decreased (Investigations) | 77 | 99
Blood potassium decreased (Investigations) | 30 | 41
Blood sodium decreased (Investigations) | 149 | 144
Blood sodium increased (Investigations) | 13 | 8
Blood triglycerides increased (Investigations) | 33 | 26
Haemoglobin decreased (Investigations) | 22 | 22
Low density lipoprotein increased (Investigations) | 124 | 93
Neutrophil count decreased (Investigations) | 62 | 78
Platelet count decreased (Investigations) | 24 | 14
White blood cell count decreased (Investigations) | 44 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 35
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Skin lesion (Skin and subcutaneous tissue disorders) | 13 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No